CLINICAL TRIAL: NCT00295113
Title: Interest of a 30 Minutes' Intermittent Work Exercise Test in Patients With Chronic Obstructive Pulmonary Disease: Cardiac and Pulmonary Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2398
Record Dates: First submitted 2005-09-13; First posted 2006-02-22 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary arterial pressure; COPD; Cardiac output; pulmonary and cardiac functions; pulmonary arterial pressure measurements
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Procedure: EFR

SUMMARY:
The aim of the study is to observe the ventilatory and cardiac function (included the pulmonary arterial pressure) during an intermittent work exercise test with high density work load.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (male and female) with moderate obstruction (FEV1/CV<60%)

Exclusion Criteria:

* acute respiratory disease
* any type of cardiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
The pulmonary arterial pressure does not increase dramatically during the 30 minutes exercise test, but decreases significantly after the first 5 minutes of exercise.

SECONDARY OUTCOMES:
The cardiac output is stable after the first 5 minutes of exercise, despite the high intensity work loads every 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg - Service des Explorations Fonctionnelles Respiratoires et de l'Exercice; Evelyne LONSDORFER-WOLF, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg - Service des Explorations Fonctionnelles Respiratoires et de l'Exercice
Locations (1):
- Hôpitaux Universitaires de Strasbourg - Service des Explorations Fonctionnelles, Strasbourg, France

REFERENCES:
- [Result] Bougault V, Lonsdorfer-Wolf E, Charloux A, Richard R, Geny B, Oswald-Mammosser M. Does thoracic bioimpedance accurately determine cardiac output in COPD patients during maximal or intermittent exercise? Chest. 2005 Apr;127(4):1122-31. doi: 10.1378/chest.127.4.1122. PMID 15821184